CLINICAL TRIAL: NCT03545165
Title: Phase I/II Dose-Escalation Trial of Combination Fractionated-dose 177Lu-J591 and 177Lu-PSMA-617 in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: 177Lu-J591 and 177Lu-PSMA-617 Combination for mCRPC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor withdrawal
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1802018988
Record Dates: First submitted 2018-05-04; First posted 2018-06-04 (Actual); Results first posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-07

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Pluvicto; gallium 68 PSMA-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- All Subjects (Experimental): 177Lu-PSMA-617 [1.85 GBq (50 mCi) - 9.25 GBq (250 mCi)] x2 doses, 2 weeks apart (Treatment Visit #1 and #2), IV administration
  177Lu-J591 [1.35 GBq/m2 or 36.5 mCi/m2] x2 doses, 2 weeks apart (Treatment Visit #1 and #2), IV administration
  68Ga-PSMA-HBED-CC [185 ±74 MBq or 5 ±2 mCi] intravenous during screening and at 12 weeks (±1 week) with standard imaging
  Interventions: Drug: 177Lu-PSMA-617; Drug: 177Lu-J591; Drug: 68Ga-PSMA-HBED-CC

INTERVENTIONS:
Drug: 177Lu-PSMA-617 — [1.85 GBq (50 mCi) - 9.25 GBq (250 mCi)]
Drug: 177Lu-J591 — [1.35 GBq/m2 or 36.5 mCi/m2]
Drug: 68Ga-PSMA-HBED-CC — [185 ±74MBq or 5 ±2 mCi]

SUMMARY:
Phase I dose escalation study with combination of 177Lu-J591 and 177Lu-PSMA-617 using a dose-fractionated regimen will be performed in patients with documented progressive metastatic CRPC. The cumulative 177Lu-J591 dose for each subject will be 2.7 GBq/m2 (73 mCi/m2) of 177Lu with 20 mg J591 and the cumulative 177Lu-PSMA-617 dose for each subject will vary (depending on the Cohort) from 3.7 GBq (100 mCi) to 18.5 GBq (500 mCi). The 177Lu-PSMA-617 dose will be escalated in up to 6 different dose levels (3+3 dose-escalation study / de-escalation design). For the phase II portion, a minimum number of 14 patients will be enrolled at MTD (including those enrolled at MTD in Phase I) and a maximum of 24.

DETAILED DESCRIPTION:
This is an open-label, single-center Phase I dose-escalation study designed to determine the dose-limiting toxicity (DLT) and the maximum tolerated dose (MTD) of combination of 177Lu-J591 and 177Lu-PSMA-617 in a two-week dose-fractionation regimen. 177Lu-J591 will be given at a moderate dose previously demonstrated to be safe x2 infusions two weeks apart. For 177Lu-PSMA-617 the dose escalation will start at 3.7 GBq (100 mCi) and escalate in increments of 1.85 GBq (50 mCi) for each dose to a planned maximum of 9.25 GBq (250 mCi) x2 doses, 2 weeks apart. Should there be unacceptable toxicity at the initial dose level, we will de-escalate to dose level -1 (1.85 GBq / 50 mCi per dose). After the phase I study has established a MTD, the Phase II, single-arm trial will start.

Patients must have documented progressive metastatic CRPC disease based on Prostate Cancer Working Group 3 (PCWG3) criteria in order to be eligible for enrollment. Upon meeting the inclusion and exclusion criteria and signing the informed consent and HIPPA form, subjects will undergo the screening. As part of the screening, subjects will get a single dose of 68Ga-PSMA-HBED-CC and will have a PET/CT. Nuclear Medicine physician(s) will review the PET/CT scans to document PSMA expression at tumor site(s).

Subjects will have Lutetium-177 Planar/SPECT Imaging on Day 8 (±1 day) after the first dose of 177Lu-J591 + 177Lu-PSMA-617. Optimal images will be performed on selected consenting subjects between the initial treatment visit #1 on Day 1 and Day 4 and prior to treatment visit #2 on D15 ±1. Subjects will be closely monitored for AEs (weekly x2 weeks, then every 2 weeks for one month, at 8 and 12 weeks, and then every 4 weeks for next 3 months).

Upon completion of investigational treatment with dose-fractionation regimen of the combination of 177Lu-J591 + 177Lu-PSMA-617, subjects will undergo 68Ga-PSMA-HBED-CC injection and same day PET/CT at the end of study visit to document treatment response. Subsequently survival data and additional treatment(s) information will be captured from their routine Standard of care (SOC) visits.

.

ELIGIBILITY:
Inclusion Criteria

1. Histologically or cytologically confirmed adenocarcinoma of prostate
2. Documented progressive metastatic CRPC based on Prostate Cancer Working Group 3 (PCWG3) criteria, which includes at least one of the following criteria:

   i. PSA progression ii. Objective radiographic progression in soft tissue iii. New bone lesions
3. ECOG performance status of 0-2
4. Have serum testosterone < 50 ng/dL. Subjects must continue primary androgen deprivation with an LHRH/GnRH analogue (agonist/antagonist) if they have not undergone bilateral orchiectomy.
5. Have previously been treated with at least one of the following:

   * Androgen receptor signaling inhibitor (such as enzalutamide)
   * CYP 17 inhibitor (such as abiraterone acetate)
6. Have previously received taxane chemotherapy, been determined to be ineligible for taxane chemotherapy by their physician, or refused taxane chemotherapy.
7. Age > 18 years
8. Patients must have normal organ and marrow function as defined below:

   * Absolute neutrophil count >2,000 cells/mm3
   * Hemoglobin ≥9 g/dL
   * Platelet count >150,000 x 109/L
   * Serum creatinine <1.5 x upper limit of normal (ULN) or calculated creatinine clearance ≥ 60 mL/min/1.73 m2 by Cockcroft-Gault
   * Serum total bilirubin<1.5 x ULN (unless due to Gilbert's syndrome in which case direct bilirubin must be normal)
   * Serum AST and ALT<1.5 x ULN in the absence of liver metastases; <3 x ULN if due to liver metastases (in both circumstances bilirubin must meet entry criteria)
9. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

1. Implantation of investigational medical device ≤4 weeks of Treatment visit #1 (Day 1) or current enrollment in oncologic investigational drug or device study
2. Use of investigational drugs ≤4 weeks or <5 half-lives of Treatment visit # 1(Day 1) or current enrollment in investigational oncology drug or device study
3. Prior systemic beta-emitting bone-seeking radioisotopes
4. Known active brain metastases or leptomeningeal disease
5. History of deep vein thrombosis and/or pulmonary embolus within 1 month of Treatment visit #1
6. Other serious illness(es) involving the cardiac, respiratory, CNS, renal, hepatic or hematological organ systems which might preclude completion of this study or interfere with determination of causality of any adverse effects experienced in this study
7. Radiation therapy for treatment of PC ≤4 weeks of Treatment visit #1
8. Patients on stable dose of bisphosphonates or denosumab, which have been started no less than 4 weeks prior to treatment start, may continue on this medication, however patients are not allowed to initiate bisphosphonate/Denosumab therapy during the DLT-assessment period of the study.
9. Having partners of childbearing potential and not willing to use a method of birth control deemed acceptable by the principle investigator and chairperson during the study and for 1 month after last study drug administration
10. Currently active other malignancy other than non-melanoma skin cancer. Patients are considered not to have "currently active" malignancy if they have completed any necessary therapy and are considered by their physician to be at less than 30% risk of relapse.
11. Known history of known myelodysplastic syndrome

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Subjects who have documented progressive metastatic CRPC disease, who meet the inclusion and exclusion criteria will be eligible for participation in this study.
Enrollment: 6 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Tagawa, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

REFERENCES:
- [Derived] Vlachostergios PJ, Niaz MJ, Skafida M, Mosallaie SA, Thomas C, Christos PJ, Osborne JR, Molina AM, Nanus DM, Bander NH, Tagawa ST. Imaging expression of prostate-specific membrane antigen and response to PSMA-targeted beta-emitting radionuclide therapies in metastatic castration-resistant prostate cancer. Prostate. 2021 Apr;81(5):279-285. doi: 10.1002/pros.24104. Epub 2021 Jan 19. PMID 33465252

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All 6 patients enrolled received both doses.
Groups:
- Cohort 1: Participants received two doses of 177Lu-J591 (60 mCi) + 177Lu-PSMA-617 (100 mCi), two weeks apart, with minimum 12 weeks of follow-up after last dose.
Period: Overall Study
Arm/Group | Cohort 1
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cohort 1
Number analyzed (Participants) | 6
Age, Continuous [Median (Full Range); unit: years] | 73 [51 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 6
Prostate specific antigen (PSA) [Median (Full Range); unit: (ng/mL)] — A tumor marker for prostate cancer (ng/mL)
  (ng/mL) | 94 [4.34 to 1398.12]
ECOG score [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) score to assess performance status; the scale ranges from 0-4 with 0 corresponding to no functional limitations; a score of 1 indicates the patient has mild limitations and may be unable to engage in physically strenuous activities
  Participants
    0 | 0
    1 | 6
Halabi (CALGB) score [Count of Participants; unit: Participants] — Halabi (Cancer and Leukemia Group B [CALGB]) score to assess prognosis in patients with metastatic prostate cancer. Three categories include low, intermediate, and high risk.
  Participants
    Intermediate | 2
    High | 4
Bone metastases [Count of Participants; unit: Participants]
  Present | 6
  Absent | 0
Lymph node metastases [Count of Participants; unit: Participants]
  Present | 4
  Absent | 2
Visceral metastases [Count of Participants; unit: Participants]
  Present | 3
  Absent | 3
Prior androgen receptor pathway inhibitor [Count of Participants; unit: Participants]
  Received | 6
  Did not receive | 0
Prior chemotherapy [Count of Participants; unit: Participants]
  Received | 5
  Did not receive | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Dose Limiting Toxicity (DLT) of Combination Therapy in a 2-Week Dose-Fractionation Regimen
Description: Dose limiting toxicity of combination therapy was determined by monitoring for adverse events following therapy
Time Frame: Approximately 3 months after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 6
Participants | 1

2. Primary Outcome: Cumulative Maximum Tolerated Dose (MTD) and/or Recommended Phase II Dose (RP2D) of Combination Therapy in a 2-Week Dose-Fractionation Regimen
Description: Cumulative maximum tolerated dose (MTD) and/or recommended phase II dose (RP2D) of combination therapy was determined by monitoring dose-limiting toxicity and adverse events in the dosing or treatment cohorts
Time Frame: Approximately 3 months after enrollment
Measure: Number; unit: mCi
Arm/Group | Cohort 1
Number analyzed (Participants) | 6
mCi | 320

3. Primary Outcome: The Proportion With PSA Decline Following the Dose-Fractionated Combination Therapy by Comparing the Change in PSA Levels After Therapy to the Baseline, Pre-Treatment PSA.
Description: The proportion of patients with PSA decline following treatment with the combination of 177Lu-J591 and 177Lu-PSMA-617 was determined by comparing PSA levels prior to and following radionuclide therapy
Time Frame: At baseline and at 2 weeks on therapy
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 6
Participants | 5

4. Secondary Outcome: Number of Subjects With Radiographic Response by RECIST 1.1 With Prostate Cancer Working Group 3 (PCWG3) Modifications
Description: Radiographic response rate was determined by scoring follow-up scans after therapy; RECIST 1.1 criteria with PCWG3 modifications were utilized
Time Frame: At the efficacy (scan) visit time point (12 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 6
Participants | 3

5. Secondary Outcome: Biochemical Progression-Free Survival by PCWG3 Criteria
Description: Biochemical progression-free survival was determined from date of first therapy to date of progression by PSA
Time Frame: Through study completion, up to 26 months
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1
Number analyzed (Participants) | 6
months | 2.5 [0 to 5]

6. Secondary Outcome: Radiographic Progression-Free Survival by PCWG3 Criteria
Description: Radiographic progression-free survival was determined from date of first treatment to date of progression on follow-up imaging
Time Frame: Through study completion, up to 26 months
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1
Number analyzed (Participants) | 6
months | 2 [0 to 6]

7. Secondary Outcome: Overall Survival Following Treatment With the Combination of 177Lu-J591 and 177Lu-PSMA-617 in a 2-Week Dose-Fractionation Regimen
Description: Overall survival following treatment with the combination of 177Lu-J591 and 177Lu-PSMA-617 was determined from date of first treatment to date of death
Time Frame: Through study completion, up to 26 months
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1
Number analyzed (Participants) | 6
months | 8 [3 to 14]

8. Secondary Outcome: Changes in CTC Count as Measured by CellSearch
Description: Patients' circulating tumor cell counts were obtained prior to and following therapy
Time Frame: At the efficacy (scan) visit time point (12 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 6
Participants
  Decline | 2
  Increase | 4

9. Secondary Outcome: Rate of Favorable CTC Count as Measured by Cell Search
Description: Patients' circulating tumor cell counts were obtained prior to and following therapy
Time Frame: At the efficacy (scan) visit time point (12 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 6
Participants | 0

10. Secondary Outcome: Rate of Favorable LDH Count
Description: Patient's LDH values were monitored prior to and following therapy
Time Frame: During treatment phase, then every 4 weeks until radiographic progression, assessed up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 6
Participants | 5

11. Other Pre Specified Outcome: Disease Assessment With PSMA-Ligand Based Imaging Prior to and Following Investigational Treatment
Description: Patients underwent Gallium-68 PSMA PET prior to investigational therapy, and lesions were scored based on SUVmax
Time Frame: Up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 6
Participants
  Highest lesion SUVmax > 5x liver SUVmean | 3
  Highest lesion SUVmax 2.5-5x liver SUVmean | 2
  Highest lesion SUVmax 1-2.5x liver SUVmean | 1

12. Other Pre Specified Outcome: Radiation Dosimetry of Combination Therapy
Description: Patients underwent SPECT following administration of radionuclides
Time Frame: Up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1
Number analyzed (Participants) | 6
Participants
  Tumor uptake at known sites of disease based on post-treatment planar imaging | 6
  No tumor uptake | 0

ADVERSE EVENTS:
Time Frame: minimum of 30 days following last dose of study drug, up to 26 months
Description: Adverse events were assessed and documented at each scheduled study visit and follow-up visit. Serious adverse events include death, life threatening adverse experiences, hospitalization or prolongation of hospitalization, disability or incapacitation, overdose, congenital anomalies and any other serious events that may jeopardize the subject or require medical or surgical intervention to prevent one of the outcomes listed in this definition.
Arm/Group | Cohort 1
All-Cause Mortality (participants affected / at risk) | 6/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=6)
dehydration (Metabolism and nutrition disorders) | 1 — The patient experienced grade 3 dehydration from vomiting, requiring hospitalization for intravenous fluids. The event was not attributed to the study drug. The event was deemed unrelated. Patient's vomiting pre-dated enrollment on the study.
back pain (Musculoskeletal and connective tissue disorders) | 1 — The patient experienced grade 3 back pain, requiring hospitalization. The adverse event was not related to the study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 (N=6)
Anorexia (Gastrointestinal disorders) | 3 — grade 1-2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 — grade 1-2
xerostomia (Gastrointestinal disorders) | 4 — grade 1-2
fatigue (General disorders) | 4 — grade 1-2
dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 — grade 1-2
transfusion reaction (General disorders) | 1 — grade 1-2
vomiting (Gastrointestinal disorders) | 1 — grade 1-2
diarrhea (Gastrointestinal disorders) | 1 — grade 1-2
hyperkalemia (Renal and urinary disorders) | 2 — grade 1-2
bruising (Skin and subcutaneous tissue disorders) | 2 — grade 1-2
hypocalcemia (Metabolism and nutrition disorders) | 2 — grade 1-2
hypokalemia (Metabolism and nutrition disorders) | 1 — grade 1-2
aspartate aminotransferase increased (Investigations) | 1 — grade 1-2
blood bilirubin increased (Investigations) | 1 — grade 1-2
creatinine increased (Investigations) | 1 — grade 1-2
nausea (Gastrointestinal disorders) | 1 — grade 1-2
hematuria (Renal and urinary disorders) | 2 — grade 3
alkaline phosphatase increased (Investigations) | 2 — grade 3
osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 — grade 3
bone pain (Musculoskeletal and connective tissue disorders) | 2 — grade 1-2
peripheral motor neuropathy (Nervous system disorders) | 1 — grade 1-2
urinary tract obstruction (Renal and urinary disorders) | 1 — grade 3
anemia (Blood and lymphatic system disorders) | 3 — grade 1-2
anemia (Blood and lymphatic system disorders) | 2 — grade 3
white blood cell decreased (Investigations) | 2 — grade 1-2
white blood cell decreased (Investigations) | 1 — grade 3
white blood cell decreased (Investigations) | 1 — grade 4
lymphocyte count decreased (Investigations) | 3 — grade 1-2
lymphocyte count decreased (Investigations) | 3 — grade 3
neutrophil count decreased (Investigations) | 3 — grade 1-2
neutrophil count decreased (Investigations) | 2 — grade 4
platelet count decreased (Investigations) | 3 — grade 1-2
platelet count decreased (Investigations) | 1 — grade 3
platelet count decreased (Investigations) | 1 — grade 4

LIMITATIONS AND CAVEATS:
The study was terminated early due to sponsor withdrawal (PSMA-617 no longer available for purchase).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/65/NCT03545165/Prot_SAP_000.pdf